CLINICAL TRIAL: NCT00521235
Title: Effects of Different Working Condition on Risk Factors in Dentists Versus Trainers. A Combined Crosssectional and Longitudinal Trial With Student and Senior Employees.
Brief Title: Effect of Different Working Conditions on Risk Factors in Dentists Versus Trainers
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University of Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Other Study IDs: ZPII-2007-10
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: risk factors; metabolic syndrome; dentists; trainers; Healthy subjects; students; seniors
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to validate the sanitary consequences of dental studies respectively the longtime executed profession. In comparison to this cohort we will also check a collective of subjects with an optimum of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 19-30 years(longitudinal)
* 55-60 years (crosssectional)
* Dentists
* Trainers

Exclusion Criteria:

* Pregnant
* CVD
* Medication; and
* Diseases affecting body composition

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: male and female students of dentistry male and female students of sports male dentists male teachers of physical education
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia S Bauer, DMD, Principal Investigator — Zahn-, Mund- und Kieferklinik, University of Erlangen-Nurnberg; Stefan Eitner, DMD, PhD, Study Director — Zahn-, Mund- und Kieferklinik, University of Erlangen; Wolfgang K Kemmler, PhD, Study Chair — University of Erlangen-Nürnberg Medical School; Simon O von Stengel, PhD, Study Chair — University of Erlangen-Nürnberg Medical School; Jürgen Weineck, PhD, MD, Study Chair — University of Erlangen-Nürnberg Medical School; Manfred Wichmann, DMD, PhD, Study Chair — Zahn-, Mund- und Kieferklinik, University of Erlangen
Locations (1):
- Zahn-, Mund- und Kieferklinik, University of Erlangen-Nurnberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Kemmler W, von Stengel S, Kohl M, Bauer J. Impact of exercise changes on body composition during the college years--a five year randomized controlled study. BMC Public Health. 2016 Jan 19;16:50. doi: 10.1186/s12889-016-2692-y. PMID 26787116